CLINICAL TRIAL: NCT00820924
Title: A Phase II Open Label, Multicenter Study to Evaluate the Efficacy and Safety of Daily Dose of Lapatinib in Advanced Breast Cancer Patients With HER-2 Non-amplified Primary Tumours and HER-2 Positive Circulating Tumour Cells or EGFR Positive Circulating Tumor Cells
Brief Title: Study of Lapatinib in Breast Cancer Patients With HER-2 Non-amplified Primary Tumors and HER-2 Positive or EGFR Positive Circulating Tumor Cells
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 105594
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Neoplasms, Breast
Keywords: HER-2; Circulating Tumour Cell (CTC); EGFR; Lapatinib (GW572016); Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LAPATINIB (Experimental): LAPATINIB 1500MG ORAL ONCE DAILY
  Interventions: Drug: LAPATINIB

INTERVENTIONS:
Drug: LAPATINIB — LAPATINIB 1500MG ORAL DOSE DAILY

SUMMARY:
The underlying biology of the various patterns of metastasis observed in different tumour types remains unclear. The detection and characterization of circulating tumour cells in cancer patients has provided important new information about the progression of metastatic events. This information has important implications for cancer prognosis and therapy.

This multicenter open-label study is designed as a two-stage three-outcome phase II trial. The aim is to evaluate the efficacy and safety of daily dose of Lapatinib in advanced breast cancer patients with HER-2 non-amplified primary tumours and HER-2 or EGFR positive circulating tumour cells. Evaluation of HER-2 and EGFR status on circulating tumour cells will be performed by the means of the CellSearch equipment (Immunicon, Huntingdon Valley, PA, USA) and FISH method (PathVysion Kit -Abbott Laboratories).

DETAILED DESCRIPTION:
Rationale: Despite recent progress in gene-expression profiling studies, the underlying biology of the various patterns of metastasis observed in different tumour types remains unclear. The detection and characterization of circulating tumour cells in cancer patients has provided important new information about the progression of metastatic events. This information has important implications for cancer prognosis and therapy.

This open label, multicenter phase II study is designed to evaluate overall tumour response rate in advanced breast cancer patients with HER-2 non amplified primary tumours with positive HER-2 or EGFR circulating tumour cells treated with the dual tyrosine kinase inhibitor GW572016 (Lapatinib).

The patients will be allocated into one of the following two strata:

Stratum 1) Italian study group: Advanced breast cancer patients with HER-2 non-amplified primary tumours and HER-2 positive circulating tumour cells Stratum 2) UK study group: Advanced breast cancer patients with HER-2 non-amplified primary tumours and EGFR positive circulating tumour cells.

All of these patients will be treated with GW572016 (Lapatinib) which targets both HER-2 or EGFR receptors. A subgroup of patients enrolled into stratum 2 will be asked to participate in an additional sub-study using Positron Emission Tomography (PET) to quantify the potential early response to lapatinib treatment.

Study Design:

This study will be a multicenter open-label, phase II study to evaluate the efficacy and safety of daily dose of Lapatinib in advanced breast cancer patients with HER-2 non amplified primary tumours and positive HER-2 or EGFR circulating tumour cells.

Patients enrolled in this study will be treated with oral Lapatinib at the dose of 1,500 mg daily on day 1 to 28 every 4 weeks (q 4 weeks).

Patients will carefully be instructed on drug administration as far as Lapatinib oral intake is concerned. A daily dose of Lapatinib is six 250 mg tablets taken approximately at the same time each day. Lapatinib must be taken either at least 1 hour before or after meal.

Dose adjustment, modification and delays are permitted according to procedures described in the protocol. Initially 16 patients in each stratum will be treated; if 1 to 3 responses are observed, 15 additional patients will be treated, up to a total of 62 subjects with 31 subjects in each stratum.

ELIGIBILITY:
Inclusion Criteria:

* Female patients at least 18 years old with HER-2 negative breast cancer.
* Patients must have evidence of HER-2 or EGFR positive circulating tumour cells in a peripheral blood sample taken at screening visit.
* Patients must have measurable, metastatic disease and no brain metastasis requiring local therapy.
* Other criteria include ECOG score 0 to 2, life expectancy > 12 weeks, baseline organ function at screening visit,
* Previous treatment with anthracyclines and/or taxanes in the neo-adjuvant, adjuvant or advanced setting, and at least one line of treatment for metastatic disease.

Exclusion Criteria:

* Unstable medical conditions, pregnant or lactating women.
* Inability to provide informed consent.
* Lack of physical integrity of the upper gastrointestinal (GI) tract.
* Co-existing malignancy or malignancies within the last 5 years with the exception of basal cell carcinoma or in-situ carcinoma, concurrent anti-cancer therapies (chemo or hormonal therapy) or investigational drugs other than study drug.
* Concurrent radiotherapy to the only target lesion or concurrent bisphosphonates if bone metastases are the only target lesions.
* Previous treatment with anti HER-2 or anti-EGFR therapies.
* Protocol specified treatment regimens that would be inappropriate for the management of the subject.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The efficacy of lapatinib in advanced breast cancer patients with HER-2 non-amplified primary tumours with HER-2 or EGFR positive circulating tumour cells. | approx. 6 mos

SECONDARY OUTCOMES:
Antitumour activity of lapatinib | approx. 6 mos
Safety of lapatinib as measured by number of AEs | approx. 6 mos
Early response of lapatinib on proliferation and the MAP kinase cascade by PET in a substudy in patients with EGFR positive CTCs only. | approx. 6 mos

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- Italy (9):
  - GSK Investigational Site, Rimini, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Bergamo, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Rozzano (MI), Lombardy
  - GSK Investigational Site, Livorno, Tuscany
  - GSK Investigational Site, Prato (PO), Tuscany
  - GSK Investigational Site, Perugia, Umbria
  - GSK Investigational Site, Ancona
- GSK Investigational Site, London, United Kingdom

REFERENCES:
- [Derived] Stebbing J, Payne R, Reise J, Frampton AE, Avery M, Woodley L, Di Leo A, Pestrin M, Krell J, Coombes RC. The efficacy of lapatinib in metastatic breast cancer with HER2 non-amplified primary tumors and EGFR positive circulating tumor cells: a proof-of-concept study. PLoS One. 2013 May 7;8(5):e62543. doi: 10.1371/journal.pone.0062543. Print 2013. PMID 23667487
- [Derived] Pestrin M, Bessi S, Puglisi F, Minisini AM, Masci G, Battelli N, Ravaioli A, Gianni L, Di Marsico R, Tondini C, Gori S, Coombes CR, Stebbing J, Biganzoli L, Buyse M, Di Leo A. Final results of a multicenter phase II clinical trial evaluating the activity of single-agent lapatinib in patients with HER2-negative metastatic breast cancer and HER2-positive circulating tumor cells. A proof-of-concept study. Breast Cancer Res Treat. 2012 Jul;134(1):283-9. doi: 10.1007/s10549-012-2045-1. Epub 2012 Apr 4. PMID 22476856